CLINICAL TRIAL: NCT06860269
Title: A 3-cohort Randomized Study Evaluating the Role of New Immunotherapeutic Agents and of Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) in Frontline Therapy of Adults With Acute Lymphoblastic Leukemia
Acronym: GRAALL-2024
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP210356
Record Dates: First submitted 2025-01-16; First posted 2025-03-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Random Allocation; blinatumomab; Drug Therapy; isatuximab; ponatinib

STUDY DESIGN:
Intervention Model Description: 3-cohort stratified multicenter multi-country prospective open-label randomized Phase III trial. In each cohort, participants will be randomized according to a 1:1 ratio (R1, R2 and R3).
  Additionnally a phase 2 single arm trial will be performed in SR patients of the Phneg BCP-ALL cohort.
  Of note, T-LL patients will be included but not randomized to receive ISA or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- GRAALL-2024/B Very High Risk - SOC (No Intervention): Phneg BCP-ALL cohort Standard of Care : ALLO HSCT
- GRAALL-2024/B High Risk - SOC (Active Comparator): Phneg BCP-ALL cohort
  Interventions: Other: Randomization 1 + Allo HSCT
- GRAALL-2024/B High risk - Blina (Experimental): Phneg BCP-ALL cohort
  Interventions: Drug: Randomization + Blinatumomab + chemotherapy
- GRAALL-2024/B Standard Risk - SOC (No Intervention): Phneg BCP-ALL cohort Standard of Care : Blinatumomab + chemotherapy
- GRAALL-2024/T - SOC (Active Comparator): T-ALL cohort
  Interventions: Other: Randomization + Standard frontline T-ALL chemotherapy backbone
- GRAALL-2024/T - Isa (Experimental): T-ALL cohort
  Interventions: Drug: Randomization + Isatuximab + Standard frontline T-ALL chemotherapy backbone
- GRAAL-2024/T - T-cell lymphoblastic lymphoma - SOC (No Intervention): Non randomized - standard care
- GRAAPH-2024 - SOC (Active Comparator): Phpos ALL cohort
  Interventions: Other: Randomization 2 + Allo HSCT
- GRAAPH-2024 - Blina/Pona (Experimental): Phpos ALL cohort
  Interventions: Drug: Randomization + Blinatumomab + Ponatinib + chemotherapy

INTERVENTIONS:
Drug: Randomization + Blinatumomab + chemotherapy — Rando 1 : BLINA will be given at 28 µg/day IVC from D1 to D28 for 2 to 4 cycles (first cycle starts with 9 µg/day for 7 days)
  Arms: GRAALL-2024/B High risk - Blina
Other: Randomization + Standard frontline T-ALL chemotherapy backbone — Rando 3 : standard of care
  Arms: GRAALL-2024/T - SOC
Drug: Randomization + Isatuximab + Standard frontline T-ALL chemotherapy backbone — Rando 3 : ISA will be given at 10 mg/kg IV for a maximum of 28 infusions starting at induction up to maintenance phase.
  Arms: GRAALL-2024/T - Isa
Drug: Randomization + Blinatumomab + Ponatinib + chemotherapy — Rando 2 :
  * PONA will be given at 45 mg/day PO during 2 cycles, 30 mg/day during 2 additional cycles, and 15 mg/day during maintenance phase or after alloHSCT
  * BLINA will be given at 28 µg/day IVC from D1 to D28 for 2 to 5 cycles (first cycle starts with 9 µg/day for 7 days). Patients allografted will receive two courses before transplant.
  Arms: GRAAPH-2024 - Blina/Pona
Other: Randomization 1 + Allo HSCT — Rando 1 : standard of care - Allogeneic Hematopoietic Stem Cell Transplantation
  Arms: GRAALL-2024/B High Risk - SOC
Other: Randomization 2 + Allo HSCT — Rando 2 : standard of care
  Arms: GRAAPH-2024 - SOC

SUMMARY:
Adult acute lymphoblastic leukemia (ALL) includes Ph-positive (Phpos) ALL, Ph-negative (Phneg) B-cell precursor (BCP) ALL and T-ALL/lymphoblastic lymphoma (LL), accounting for approximately 25, 50 and 25% of all cases, respectively. In younger adults, the results associated with standard therapy have markedly improved in these 3 groups, due to chemotherapy intensification in the BCP and T groups and addition of TKIs in the Phpos group, respectively. This led to reevaluate the role of allogeneic hematopoietic stem cell transplantation (HSCT) in first remission, which is generally now indicated only in higher-risk patients, mostly defined as those with persistent high levels of minimal residual disease (MRD). Nevertheless, event-free survival (EFS) remains at 60-70% at 3 years, meaning there is still room for further improvements.

Fortunately, new immunotherapies have been approved to treat relapsed/refractory (R/R) BCP-ALL patients, including the anti-CD19 bispecific T-cell engager blinatumomab (BLINA, Blincyto®, Amgen). 4 BLINA is also approved for the frontline treatment of patients with persistent high measurable residual disease (MRD) levels after initial therapy (IG/TR MRD ≥0.1% (≥1.10-3

)). BLINA has been also evaluated frontline in combination with TKI in the Phpos group leading to promising outcome improvements. Toxicities associated with these combined treatments seem to be limited and manageable. In the Phpos ALL subset, the third-generation tyrosine kinase inhibitor ponatinib (PONA, Iclusig®, Incyte) has also been evaluated frontline with promising results when compared to 1st or even 2nd generation TKI. In the T-ALL/LL subset, anti-CD38 antibodies, approved to treat patients with multiple myeloma, are potential drugs of interest. The anti-CD38 antibody isatuximab (ISA, Sarclisa®, Immunogen, Sanofi-Aventis) is currently approved to treat myeloma patients in 2nd line. In vitro and in vivo preclinical studies suggest that CD38 is a relevant target in T-ALL and that isatuximab may be useful to eradicate residual disease in this subgroup of patients. Incorporation/combination of these new agents into frontline adult ALL therapy could allow reducing relapse incidence and prolonging survival in these patients, challenging the indication for HSCT in first complete remission (CR).

The present GRAALL-2024 study is a prospective multicenter multi-country 3-cohort randomized clinical trial.

The 3 cohorts are :

GRAALL-2024/B : Phneg BCP-ALL GRAAPH-2024 : Phpos ALL GRAALL-2024/T : T-ALL/LL

Eligible patients will be allocated to one on the 3 study cohorts during a common treatment prephase. The primary objective of the study is to improve the outcome of younger adults with ALL through optimal frontline incorporation of new antibody-based therapies, including BLINA in Phneg/pos BCP-ALL patients and ISA in T-ALL/LL patients, and to refine indication for allogeneic HSCT in first remission in Phneg/pos BCP-ALL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 65 years old
2. Newly diagnosed ALL or T-LL according to the WHO criteria
3. Immunophenotypic, cytogenetic and/or FISH and molecular evaluation performed and allowing classifying the patient in one of the Phpos ALL, Phneg BCP-ALL or T-ALL/LL cohorts
4. Not previously treated except with corticosteroids and/or intrathecal therapy (prephase)
5. Eligible for allo-HSCT if Phpos ALL or Phneg BCP-ALL
6. ECOG performance status ≤2
7. Patient willing and able to understand the protocol requirements and comply with the treatment schedule, scheduled visits, electronic patient outcome reporting, exams and other requirements of the study
8. Patients has signed written inform consent
9. Willingness of women of child-bearing potential (WOCBP) and male subjects whose sexual partners are WOCBP to use an effective form of contraception, i.e. methods with a failure rate of <1% per year when used consistently and correctly, during the study and at least 6 months thereafter
10. Eligible for National Health Insurance (for French patients)

Exclusion Criteria:

Common exclusion criteria :

1. Patient previously treated with systemic chemotherapy, antibody-based therapy or TKI
2. Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention
3. History or presence of clinically relevant CNS pathology such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, coordination/movement disorder, autoimmune disease with CNS involvement, psychosis (with the exception of CNS leukemia that is well controlled with intrathecal therapy)
4. Patients with LVEF<50% or other clinically significant heart disease (e.g. unstable angina, congestive heart failure, uncontrolled hypertension)
5. Prior documented chronic liver disease. Inadequate hepatic functions defined as AST or ALT > 5 x the institutional upper limit of normal (ULN), or > 5 x ULN unless if considered due to leukemia. Total bilirubin > 1.5 x ULN unless if considered due to leukemia or Gilbert/Meulengracht
6. Estimated glomerular filtration rate (GFR) < 50 mL/mn using the MDRD equation
7. Chronic pancreatitis or acute pancreatitis within 6 months before study start
8. Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory) or active infection with Hepatitis B or C.
9. Concurrent severe diseases which exclude the administration of therapy
10. Treatment with any other investigational agent or participating in another trial within 30 days prior to entering this study
11. Pregnancy and breast feeding
12. Patients unwilling or unable to comply with the protocol
13. Patients under a legal protection regime (guardianship, trusteeship, judicial safeguard)
14. Chronic or current active uncontrolled infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment
15. Current use of prohibited medication
16. Known hypersensitivity or severe reaction to ponatinib (GRAAPH), blinatumomab (GRAAPH and GRAALL-B) , isatuximab (GRAALL-T) or their excipients.
17. Receipt of live (including attenuated) vaccines or anticipation of need for such vaccines during the study

If patients with Phpos ALL:

1. Complete left bundle branch block, right bundle branch block plus left anterior hemiblock, bi-fascicular block
2. History of or presence of clinically significant ventricular or atrial tachyarrhythmias
3. Clinically significant resting bradycardia (< 50 beats per minute)
4. Congenital long QT syndrome or QTcF > 470 msec on screening ECG. If QTc > 470 msec and electrolytes are not within normal ranges before ponatinib dosing, electrolytes should be corrected and then the patient rescreened for QTcF criterion
5. Currently taking drug(s) that are known to have a risk of causing prolonged QTc or TdP unless the drug(s) can be changed to acceptable alternatives (ie, an alternate class of agents that do not affect the cardiac conduction system), or the participant can safely discontinue the drug(s)
6. Previous myocardial infarction within the last 12 months
7. Symptomatic peripheral vascular disease
8. History of ischemic stroke or transient ischemic attacks (TIAs) within the last 12 months
9. Significant bleeding disorder or thrombophilia unrelated to the underlying malignancy indication for study participation
10. Gastrointestinal disorders, such as malabsorption syndrome or any other illness that could affect oral absorption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2035-03-15 (Estimated); Study Completion 2035-03-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival | At 5 years
  For GRAAL-2024/B HR patients (phase 3)
Overall survival | At 5 years
  For GRAAL-2024/B SR patients (phase 2)
Event-Free Survival | At 5 years
  For GRAAL-2024/T patients (phase 3)
Overall survival | At 5 years
  For GRAAPH-2024 patients (phase 3) - Phpos ALL

SECONDARY OUTCOMES:
Overall survival | At 5 years
  in the T-ALL/LL cohorts
Event Free Survival | At 5 years
Relapse Free Survival | At 5 years
Hematological complete response rate | At 45 days
  After induction
Hematological complete response rate | At 4 months
  After consolidation
Measurable residual disease (MRD) response level | At inclusion
  (IG/TR and BCR::ABL1 markers) at diagnosis
Measurable residual disease (MRD) response level - non graft patients | Up to 6 months
  (IG/TR and BCR::ABL1 markers) After each treatment cycle until maintenance (4 to 5 times)
Measurable residual disease (MRD) response level - graft patients | Through study completion, approximately 5 years
  (IG/TR and BCR::ABL1 markers) At day 100 post-HSCT and every 3 months post HSCT for patients receiving allo-HSCT during maintenance up to 2 years
Measurable residual disease (MRD) response level | Up to 5 years
  (IG/TR and BCR::ABL1 markers) At relapse
Early mortality | At day 30
Early mortality | At day 60
Early mortality | At day 90
Cumulative incidence of relapse (CIR) | At 5 years
Cumulative incidence of non relapse mortality | At 5 years
Transplant-related mortality (TRM) | At 5 years
  For graft patients
Graft-versus-host-disease (GvHD) incidence | At 5 years
  For graft patients
Number of patients who experience one or more Adverse Event (AEs) or Serious Adverse Event (SAEs) | At 5 years
Rate of patients who experience one or more Adverse Event (AEs) or Serious Adverse Event (SAEs) | At 5 years
Quality of life level | Until 5 years
  Assessed with EQ5D 5L It evaluates five dimensions : mobility, self-care, usual activities, pain/discomfort and anxiety/depression and each dimension has five levels : no problems, slight problems, moderate problems, severe problems and extreme problems. Answers are given on a 5-point scale by domain, the higher the score, the poorer the quality of life.
  At each study visit
Incremental cost effectiveness and cost utility ratio | At 5 years
  Defined as the difference in total costs divided by the difference in survival and in quality adjusted life years

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint Louis, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided